CLINICAL TRIAL: NCT01286168
Title: Trial of Drain Antisepsis After Tissue Expander Breast Reconstruction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: University of California, San Francisco (Other); Ethicon, Inc. (Industry)
Responsible Party: Principal Investigator, Amy C. Degnim, MD, Mayo Clinic
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 10-008061; UL1TR000135 (NIH)
Record Dates: First submitted 2011-01-26; First posted 2011-01-31 (Estimated); Results first posted 2014-10-20 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Nonmalignant Breast Conditions; Breast Cancer
Keywords: Bilateral breast mastectomy; Immediate tissue expanders reconstruction
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antisepsis Side (Experimental): A chlorhexidine gluconate disk (BioPatch) covered by an occlusive adhesive dressing (Tegaderm) will be applied to the intervention drain sites and changed every three days. The drainage bulb will be irrigated with 10ml of 0.125% sodium hypochlorite (Dakin's solution) twice a day.
  Interventions: Device: Sodium hypochlorite (Dakin's Solution); Device: Chlorhexidine gluconate disk; Device: Occlusive Adhesive Dressing
- Control Side (Other): Standard drain care will be performed twice a day or three times if bulb is full and needs to be emptied. Standard drain care consists of stripping the tubing, emptying the drainage bulb, recording the volume of fluid, and cleaning the drain site with a cotton swab dipped in rubbing alcohol. The drain exit will be covered with a dry sterile gauze dressing and changed after each episode of drain care.
  Interventions: Procedure: Control

INTERVENTIONS:
Device: Sodium hypochlorite (Dakin's Solution) — 10 ml of 0.125% sodium hypochlorite (Dakin's solution) irrigation to the drainage bulb two times a day
  Other Names: Dakin's solution; Wound cleanser
  Arms: Antisepsis Side
Device: Chlorhexidine gluconate disk — Apply one chlorhexidine disk to the intervention drain site(s) and change every three days
  Other Names: BioPatch Protective Disk with CHG
  Arms: Antisepsis Side
Procedure: Control — Standard drain care will be performed twice a day or three times if bulb is full and needs to be emptied. Standard drain care consists of stripping the tubing, emptying the drainage bulb, recording the volume of fluid, and cleaning the drain site with a cotton swab dipped in rubbing alcohol. The drain exit will be covered with a dry sterile gauze dressing and changed after each episode of drain care.
  Arms: Control Side
Device: Occlusive Adhesive Dressing — A chlorhexidine gluconate disk (BioPatch) covered by an occlusive adhesive dressing (Tegaderm) will be applied to the intervention drain sites and changed every three days.
  Other Names: Tegaderm CHG Dressing
  Arms: Antisepsis Side

SUMMARY:
Surgical site infection (SSI) after breast and axillary surgery occurs more often than for other clean surgical procedures. Infection in the setting of a tissue expander can be devastating and can lead to early implant loss and failed reconstruction. Surgical drains have been noted as a potential source for surgical site infections. Hypothesis: Bacteria present in surgical drains after tissue expander reconstruction may be decreased by simple and inexpensive local antiseptic interventions.

DETAILED DESCRIPTION:
Surgical Site infection after breast surgical procedures occurs more frequently than for other clean surgical procedures. Considering the large numbers of patients who undergo breast-related procedures per year and the increasing use of immediate breast reconstruction with placement of tissue expanders or immediate implant reconstruction, a surgical site infection involving the implant can result in its removal and a failed reconstruction.

The primary aim of the study is to determine if chlorhexidine disk application and irrigation of the drainage bulb with dilute Dakin's solution (buffered sodium hypochlorite solution)after tissue expander breast reconstruction or immediate implant reconstruction, effectively decreases rates of bacterial colonization in drain fluid compared to standard care.

Methods:

Patients undergoing bilateral immediate reconstruction with tissue expander placement will have one surgical site treated with standard drain care and the other treated with a drain antisepsis regimen. Drain antisepsis intervention will consist of two measures: 1) placement of a chlorhexidine sponge dressing at the drain exit site, and 2) twice daily irrigation of the drainage bulb with dilute Dakin's solution (buffered hypochlorite).

All patients will undergo semiquantitative cultures of the drain bulb at one week postoperatively. This culture will be repeated at the time of drain removal, with simultaneous cultures of the fluid in the bulb as well as an internal segment of each removed drainage tube. All patients will be evaluated for clinical signs of infection and for any adverse reactions to the drain antisepsis at the follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Females or males age 18-90 able to give informed consent
* Undergoing bilateral mastectomy with immediate expander reconstruction or immediate implant reconstruction
* May have either malignant or benign breast condition

Exclusion Criteria:

* Antibiotic use in the fourteen days prior to surgical date
* Undergoing unilateral tissue expander reconstruction
* Documented allergy to chlorhexidine gluconate
* Prior radiation therapy to the breast or chest wall (ie for breast conservation or mantle radiation for Hodgkin's disease)
* Documented allergy to all three of the following antibiotics: cephalosporin, trimethoprim/sulfamethoxazole, and levofloxacin
* Pregnant women
* Vulnerable subjects - prisoners, institutionalized individuals
* Non-English speaking patients without adequate interpreter assistance

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2011-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy C Degnim, M.D., Principal Investigator — Mayo Clinic, Rochester, MN
Locations (2):
- United States (2):
  - UCSF, San Francisco, California
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- [Derived] Degnim AC, Scow JS, Hoskin TL, Miller JP, Loprinzi M, Boughey JC, Jakub JW, Throckmorton A, Patel R, Baddour LM. Randomized controlled trial to reduce bacterial colonization of surgical drains after breast and axillary operations. Ann Surg. 2013 Aug;258(2):240-7. doi: 10.1097/SLA.0b013e31828c0b85. PMID 23518704

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at the Mayo Clinic, Rochester, Minnesota, and the University of California, San Francisco, California. Eligible subjects were recruited prospectively from the breast surgical practices between May 2011 and June 2013.
Pre-assignment Details: Six subjects did not start study therapy: One subject became a screen failure when her procedure was changed to a lumpectomy. For one subject, no Dakin's solution was available at the pharmacy. Four subjects withdrew, changing their minds about participating.
Groups:
- Entire Study Population: Because a paired study design was used (only bilateral procedures), each subject served as her own control. Randomization assigned which side (right or left) would receive the antisepsis interventions, and the contralateral side received standard drain care.
Period: Overall Study
Arm/Group | Entire Study Population
Started | 104
Completed | 101
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Surgical Drains Fell Out at Home | 2

BASELINE CHARACTERISTICS:
Population: This number includes all subjects who started study therapy.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 104
Age, Continuous [Median (Full Range); unit: years] | 46 [25 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 104
Body Mass Index [Median (Full Range); unit: kg/m^2] — Body Mass Index (BMI) is a health index for comparing weight to height. BMI is a person's weight in kilograms (kg) divided by his or her height in meters squared. The body mass index is an indication if a person is at a suitable weight for his height on an approximation of body fat. A body mass index of under 20 is considered to be underweight, while a body mass index between 20 to 25 is considered healthy. A body mass index in the range of 25 to 30 is regarded as overweight. A body mass index over 30 is regarded as obese.
  kg/m^2 | 23.8 [17 to 45.1]
American Society of Anesthesiologists (ASA) Class [Number; unit: participants] — The ASA physical status classification system is a system for assessing the fitness of cases before surgery. Class 1: Healthy person. Class 2: Mild systemic disease. Class 3: Severe systemic disease. Class 4: Severe systemic disease that is a constant threat to life. Class 5: A moribund person who is not expected to survive without the operation. Class 6: A declared brain-dead person whose organs are being removed for donor purposes.
  participants
    Class I | 19
    Class II | 77
    Class III | 8
Operative Time [Median (Full Range); unit: hours] | 5.1 [2.9 to 9.3]
Smoking within 4 weeks preoperation [Number; unit: participants]
  Yes | 4
  No | 99
  Unknown | 1
Diagnosis of diabetes [Number; unit: participants]
  Yes | 3
  No | 101
Neoadjuvant chemotherapy [Number; unit: participants]
  Yes | 32
  No | 72
Indication for surgery [Number; unit: participants] — Contralateral prophylactic mastectomy (CPM)
  participants
    Unilateral cancer with CPM | 72
    Bilateral prophylactic mastectomy | 24
    Bilateral cancer | 8
Type of Preoperative Antibiotic [Number; unit: participants]
  Cefazolin | 92
  Clindamycin | 6
  Levofloxacin | 3
  Vancomycin | 3
Type of Operation (Antisepsis side) [Number; unit: participants]
  Mastectomy only | 58
  Mastectomy + sentinel lymph node biopsy (SLNB) | 35
  Mastectomy + axillary lymph node dissection (ALND) | 11
Type of Operation (Control Side) [Number; unit: participants]
  Mastectomy only | 61
  Mastectomy + sentinel lymph node biopsy (SLNB) | 32
  Mastectomy + axillary lymph node dissection (ALND) | 11
Type of Mastectomy (Antisepsis Side) [Number; unit: participants]
  Skin-sparing | 37
  Nipple-sparing | 67
Type of Mastectomy (Control Side) [Number; unit: participants]
  Skin-sparing | 36
  Nipple-sparing | 68
Indication for Mastectomy (Antisepsis Side) [Number; unit: participants]
  Cancer | 46
  Risk-reducing | 58
Indication for Mastectomy (Control Side) [Number; unit: participants]
  Cancer | 42
  Risk-reducing | 62
Number of Drains (Antisepsis Side) [Number; unit: participants]
  1 | 52
  2 | 47
  3 | 5
Number of Drains (Control Side) [Number; unit: participants]
  1 | 54
  2 | 42
  3 | 8
Type of Reconstruction (Antisepsis Side) [Number; unit: participants]
  Tissue expander | 95
  Direct-to-implant | 9
Type of Reconstruction (Control Side) [Number; unit: participants]
  Tissue expander | 95
  Direct-to-implant | 9
Acellular dermal matrix used (Antisepsis Side) [Number; unit: participants]
  Yes | 75
  No | 29
Acellular dermal matrix used (Control Side) [Number; unit: participants]
  Yes | 76
  No | 28
Intraoperative Fill Volume (Antisepsis Side) [Median (Full Range); unit: mL] — Interoperative fill volume available in n=101 participants, and missing in n=3 participants.
  mL | 150 [0 to 800]
Intraoperative Fill Volume (Control Side) [Median (Full Range); unit: mL] — Interoperative fill volume available in n=101 participants, and missing in n=3 participants.
  mL | 150 [0 to 800]
Number of Lymph Nodes Removed (Antisepsis Side) [Median (Full Range); unit: lymph nodes] — Among sides with either sentinel lymph node biopsy (SLNB) or axillary lymph node dissection (ALND), n=46 antisepsis side.
  lymph nodes | 3 [1 to 33]
Number of Lymph Nodes Removed (Control Side) [Median (Full Range); unit: lymph nodes] — Among sides with either SLNB or ALND, n=43 control.
  lymph nodes | 4 [1 to 36]
Maximum Drain Duration (Antisepsis Side) [Median (Full Range); unit: days] — Maximum duration across all drains on a given side.
  days | 13 [6 to 50]
Maximum Drain Duration (Control Side) [Median (Full Range); unit: days] — Maximum duration across all drains on a given side.
  days | 13 [6 to 34]
Adjuvant Radiation Therapy (Antisepsis Side) [Number; unit: participants] — Adjuvant radiation therapy within one year, but prior to tissue expander exchange.
  participants
    Yes | 7
    No | 97
Adjuvant Radiation Therapy (Control Side) [Number; unit: participants] — Adjuvant radiation therapy within one year, but prior to tissue expander exchange.
  participants
    Yes | 8
    No | 96

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Drain Bulb Fluid Bacterial Colonization at Approximately 1 Week
Description: Bacterial growth was defined as plate growth of 1+ or greater. Drains were removed at variable times across patients, per clinical indication. When clinically indicated, some patients did have their drains removed at the one week visit, in which case they only had one bulb fluid culture.
Time Frame: Approximately 1 week after surgery
Population: Analysis was modified intent-to-treat (IIT); subjects who withdrew or were screen failures before study intervention were excluded. All patients who completed were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Entire Study Population
Number analyzed (Participants) | 101
participants
  Antisepsis Side | 10
  Control Side | 21
Statistical Analysis 1: Comparison: Entire Study Population; Antisepsis and Control sides were compared; Test type: Superiority or Other; p = 0.02, McNemar

2. Secondary Outcome: Number of Subjects With Drain Tubing Colonization at Removal
Description: Drain tubing colonization was defined as greater than 50 colony forming units. Drains were removed at variable timepoints based on the clinical situation.
Time Frame: Approximately two weeks after surgery
Population: Analysis was modified intent-to-treat; subjects who withdrew or were screen failures before study intervention were excluded. All patients who completed were included in the analysis. 2 subjects missed endpoint due of protocol deviation or discontinuation, and 2 had the sterility of their drain tubing compromised by external exposures.
Measure: Number; unit: participants
Arm/Group | Entire Study Population
Number analyzed (Participants) | 97
participants
  Antisepsis Side | 0
  Control Side | 6
Statistical Analysis 1: Comparison: Entire Study Population; Antisepsis and Control sides were compared; Test type: Superiority or Other; p = 0.03, McNemar

3. Secondary Outcome: Number of Subjects With Drain Bulb Fluid Bacterial Colonization at Removal
Description: Bacterial growth was defined as plate growth of 1+ or greater. Drains were removed a variable times across patients, per clinical indication. A second bulb culture was obtained later than 1 week ONLY in those drains that were not removed at 1 week.
Time Frame: Approximately 2 weeks after surgery
Population: Analysis was modified intent-to-treat (IIT). Reported here only in those subjects where drain removal was later than primary endpoint collection.
Measure: Number; unit: participants
Arm/Group | Entire Study Population
Number analyzed (Participants) | 72
participants
  Antisepsis Side | 14
  Control Side | 28
Statistical Analysis 1: Comparison: Entire Study Population; Antisepsis and Control sides were compared; Test type: Superiority or Other; p = 0.003, McNemar

4. Secondary Outcome: Number of Subjects With Surgical Site Infection Within 30 Days
Time Frame: Approximately 30 days after surgery
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Entire Study Population
Number analyzed (Participants) | 104
participants
  Antisepsis Side | 0
  Control Side | 4
Statistical Analysis 1: Comparison: Entire Study Population; Antisepsis and Control sides were compared; Test type: Superiority or Other; p = 0.13, McNemar

5. Secondary Outcome: Number of Subjects With Surgical Site Infection Within 1 Year
Time Frame: Approximately one year after surgery
Measure: Number; unit: participants
Arm/Group | Entire Study Population
Number analyzed (Participants) | 104
participants
  Antisepsis Side | 3
  Control Side | 6
Statistical Analysis 1: Comparison: Entire Study Population; Antisepsis and Control sides were compared; Test type: Superiority or Other; p = 0.45, McNemar

6. Primary Outcome: Per Drain Analysis: Drain Bulb Fluid Colonization at Approximately 1 Week
Time Frame: Approximately 1 week after surgery
Population: as for outcome 1
Measure: Number; unit: drains
Units Other Than Participants: drains
Arm/Group | Entire Study Population
Number analyzed (Participants) | 101
Number analyzed (drains) | 317
drains
  Antisepsis side n=157 drains | 11
  Control side n=160 drains | 25
Statistical Analysis 1: Comparison: Entire Study Population; Antisepsis and Control sides were compared. Unadjusted p-value from generalized linear mixed effect model accounting for correlation among multiple drains from the same patient; Test type: Superiority or Other; p = 0.02, Mixed Models Analysis
Statistical Analysis 2: Comparison: Entire Study Population; Antisepsis and Control sides were compared. P-value from generalized linear mixed effect model accounting for correlation among multiple drains from the same patient. P-value was adjusted for side- and drain-specific variables: indication (cancer or prophylaxis), operation (mastectomy only, mastectomy+SLNB, mastectomy +ALND), and drain duration; Test type: Superiority or Other; p = 0.02, Mixed Models Analysis

7. Secondary Outcome: Per Drain Analysis: Drain Tubing Colonization at Removal
Time Frame: Approximately one month after surgery
Population: as for outcome 2
Measure: Number; unit: drains
Units Other Than Participants: drains
Arm/Group | Entire Study Population
Number analyzed (Participants) | 97
Number analyzed (drains) | 305
drains
  Antisepsis side, n=151 drains | 0
  Control side, n=154 | 6
Statistical Analysis 1: Comparison: Entire Study Population; Antisepsis and Control sides were compared. Due to zero events in the antisepsis side for this endpoint, p-value was derived from likelihood-ratio test comparing the intercept only model to the model with intercept and treatment side included; Test type: Superiority or Other; p = 0.004, Likelihood-ratio test

8. Secondary Outcome: Per Drain Analysis: Drain Bulb Fluid Colonization at Removal
Time Frame: Approximately one month after surgery
Population: as for outcome 3
Measure: Number; unit: drains
Units Other Than Participants: drains
Arm/Group | Entire Study Population
Number analyzed (Participants) | 72
Number analyzed (drains) | 173
drains
  Antisepsis side, n=85 drains | 14
  Control side, n=88 drains | 33
Statistical Analysis 1: Comparison: Entire Study Population; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis
Statistical Analysis 2: Comparison: Entire Study Population; [analysis description as in outcome 6, analysis 2]; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Eligible subjects were recruited prospectively from the breast surgical practices between May 2011 and June 2013.
Description: All subjects underwent a mandatory follow-up visit approximately one week after surgery, at which time surgical sites are evaluated and appropriate study cultures obtained. Additional visits were made for clinical care; follow up phone calls were also made to the subjects.
Arm/Group | Antisepsis Side | Control Side
Serious Adverse Events (participants affected / at risk) | 0/104 | 0/104
Other Adverse Events (participants affected / at risk) | 3/104 | 6/104
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Antisepsis Side (N=104) | Control Side (N=104)
Surgical Site Infection (Infections and infestations) | 3 | 6 — Surgical site infection per operated side within one year of operation. Includes only infections that occurred before a secondary operation such as tissue expander/implant exchange.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No